CLINICAL TRIAL: NCT06043141
Title: Investigation of the Relationship Between Pain Sensitization and Ultrasonographic and Electrodiagnostic Parameters in Carpal Tunnel Syndrome
Brief Title: Investigation of the Relationship Between Pain Sensitization and Diagnostic Parameters in Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Feyza Nur Yucel, Specialist, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: 23-517
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Central Sensitisation; Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with carpal tunnel syndrome: Patients with carpal tunnel syndrome
  Interventions: Diagnostic Test: Nerve ultrasound; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Pressure pain threshold
- Control group: Healthy control
  Interventions: Diagnostic Test: Nerve ultrasound; Diagnostic Test: Pressure pain threshold

INTERVENTIONS:
Diagnostic Test: Nerve ultrasound — Ultrasonographic evaluation of the median nerve at the carpal tunnel and adjacent levels
Diagnostic Test: Nerve conduction studies — Upper extremity nerve conduction studies including median-ulnar sensory and motor responses
  Groups: Patients with carpal tunnel syndrome
Diagnostic Test: Pressure pain threshold — Pain pressure threshold (PPT) is used to measure deep muscular tissue pain sensitivity.
  Other Names: PPT

SUMMARY:
The aim of this observational, cross-sectional study is to investigate the relationship between pain sensitization and ultrasonographic and nerve conduction studies in patients diagnosed with carpal tunnel syndrome (CTS).

The main questions it aims to answer are:

* Can threshold values be determined ultrasonographically and electrodiagnostically in patients who develop pain sensitization?
* Are pressure pain threshold values and central sensitization inventory scores correlated with ultrasonographic and nerve conduction studies of the median nerve?

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common nerve entrapment and the main mechanism is compression of the median nerve under the transverse ligament at the wrist level. Its incidence varies between 6.3-11.7% in the general population. In CTS, neuropathic complaints such as numbness, burning and tingling in the palmar face of the first two fingers, which are the innervation area of the median nerve, and fatigue in the hand are the most common symptoms. However, it has been reported that these complaints in most patients are not limited to the innervation area of the median nerve but also spread to other neighboring areas. This has been found to be associated with the development of central sensitization in CTS patients, and extra-median symptoms are suggested to be a clinical marker of pain sensitization. The term central sensitization is explained as an increase in pain sensitivity due to the amplification of neuron-derived signals in the central nervous system.Research shows that ongoing damage to the median nerve stimulates neurons located in the central nervous system, advancing the central sensitization process. Although the diagnosis of CTS is made electrodiagnostically with typical clinical findings, in recent years ultrasound has been frequently used in the diagnosis of CTS because it is non-invasive, fast and reliable. Cross-sectional area and echogenicity of the median nerve are the most frequently evaluated parameters at the carpal tunnel with ultrasound. Studies focus on the clinical relationship of central sensitization in CTS, but its relationship with ultrasonographic and electrodiagnostic data is not yet known.Based on this, this study aimed to investigate the relationship between pain sensitization and electrodiagnostic and ultrasonographic parameters in patients diagnosed with CTS.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with carpal tunnel syndrome based on clinical and electrodiagnostic findings
* Agreeing to participate in the study

Exclusion Criteria:

* Concomitant history of diabetes, systemic inflammatory disease, active infection and malignancy
* Having a disease with neuropathic pain such as polyneuropathy, radiculopathy,multiple sclerosis
* Not agreeing to participate in the study
* History of surgery due to CTS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CTS
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Pressure pian threshold | 3 months
  Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. Algometer is used in the measurement and low values are interpreted in favor of increased sensitivity.

SECONDARY OUTCOMES:
Central sensitization inventory (CSI) | 3 months
  Clinical instrument used in the diagnosis of central sensitization. A CSI part-A score of 40 and above is significant in the diagnosis.
hand grip strength | 3 months
  Grip strength is a measure of muscle strength or the maximum force/tension produced by one's forearm muscles and is measured with a hand dynamometer.
Visual analog scale | 3 months
  The visual analog scale (VAS) is a validated subjective measure for pain, scored in the 0-10 range (0:no pain; 10: worst pain).
Upper extremity nerve conduction studies | 3 months
  Latency, conduction velocity and amplitude values obtained in bilateral median-ulnar motor and sensory nerve conduction studies.
median nerve ultrasound | 3 months
  Median nerve cross-sectional area and echogenicity measurement
Short form-12 | 3 months
  The 12-item Short Form Questionnaire (SF-12) is used for objective measurement of quality of life. Low scores are associated with poor in quality of life.
Self Leeds Assessment of Neuropathic Symptoms and Sign (S-LANSS) | 3 months
  S-LANSS is a 7-question scale used to define pain of neuropathic origin and a score of 12 points or more is in favor of the presence of neuropathic pain.
Boston Carpal Tunnel Questionnaire (BCTQ) | 3 months
  The Boston Carpal Tunnel Score is a patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome. Two subscores are calculated: Symptom Severity Scale (SSS) and Functional Status Scale (FSS); higher scores indicate worse symptoms or function.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Asst.Prof, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Sultan Abdülhamid Han Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Dataset sharing is not planned